CLINICAL TRIAL: NCT04576221
Title: Comparative Study Between NIV With Using CPAP Mask Versus Stacked Breathing on Chest Expansion and Pulmonary Function in Patient With Pneumonia
Brief Title: Comparative Study Between CPAP Mask and Stacked Breathing o Pneumonia
Acronym: CPAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ahmed talaat ahmed aly (Other)
Collaborators: Ain Shams University (Other)
Responsible Party: Sponsor-Investigator, Ahmed talaat ahmed aly, clinical professor, Assiut University
Organization: Assiut University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: stacked breathing
Record Dates: First submitted 2020-08-31; First posted 2020-10-06 (Actual); Last update posted 2020-10-06 (Actual); Status verified 2020-10

CONDITIONS: Pulmonary Function
Keywords: stacked breathing; CPAP mask; pneumonia
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Intervention Model Description: use of two manner of breathing for patients with pneumonia.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- stacked breathing group (Experimental): experimental group received staked breathing exercise for 7 days , 3 sessions per day, 7-8 times per session
  Interventions: Device: stacked breathing exercise
- CPAP group (Experimental): experimental group received NIV with CPAP mask
  Interventions: Device: NIV by CPAP mask

INTERVENTIONS:
Device: stacked breathing exercise — • Breath stacking was done using a "bag" which is a simple device used to give artificial breaths..
  * It is best done in a sitting position but can be done reclining or lying flat whichever position is used, try to avoid slouching. If sitting: rest against the back of a chair and keep the shoulders, arms and hands relaxed.
  * If using the mouthpiece, place the lips tightly around the mouthpiece to create a tight seal.
  Arms: stacked breathing group
Device: NIV by CPAP mask — provides pressurized air through a mask to help push air into your lungs and help you breathe
  Arms: CPAP group

SUMMARY:
the study aimed to compare the effect of using NIV with using CPAP mask and stacked breathing exercise and its efficacy on chest expansion and pulmonary functions in pneumonic patients.

DETAILED DESCRIPTION:
Introduction Pneumonia represents a frequent complication in patients in ICU with rates up to 56% . Although oxygen therapy is the cornerstone for pneumonia treatment, its efficacy might be minimized because of shunt effects due to the presence of pulmonary exudate and atelectasis. To improve oxygenation, alveolar recruitment obtained through the application of either invasive or non-invasive mechanical ventilation (NIV) might be necessary, especially in severe pneumonia .

The role of NIV as a tool to treat pneumonia has dramatically increased over the past decades and its efficacy has been well studied in clinical practice, especially in treating acute cardiogenic pulmonary edema and exacerbation of Chronic Obstructive Pulmonary Disease (COPD). Concerning NIV treatment in patients with pneumonia, its use has been proved to be effective only in patients with COPD and in immunocompromised patients with lung infiltrates . The lack of strong evidence in literature led international experts to suggest only cautious trials of NIV in well-selected patients with pneumonia and in trained settings with a clear caveat to avoid a delay in endotracheal intubation . One method of NIV is Continuous Positive Airway Pressure (CPAP) which is used to administer fresh gas pressure to the spontaneously breathing patient. By opening more alveolar spaces, CPAP increases the number of functional airways, thereby reducing total resistance. The success of CPAP therapy is highly influenced by patient compliance and the level of comfort provided by the CPAP mask and headgear. If the patient is able to tolerate CPAP and use it correctly, its effective rate is nearly 100% . The majority of patients fail the treatment not because of its low efficacy for maintaining upper airway patency but because of intolerance .

There are different types of physiotherapy exercises which can benefit patient with pneumonia and help lung recruitment as CPAP ventilation but it is more tolerance to patient than use of CPAP mask . one of these exercises is breathing stacking which is a breathing exercise to help improve and maintain the size of breath that the patient is able to take and can be used regularly to help the patient clear mucus from his chest (secretion clearance).

It can also be used to help improve the strength of the cough and voice . It is mainly used for people with weak breathing muscles which makes breathing and coughing difficult. Patients with neuromuscular diseases often have weakness of their breathing (respiratory) muscles which affects how well the respiratory system works. It is also used for people with bone or structural problems which cause a small / altered chest shape making coughing difficult .

The aim of this study is to compare the effect of NIV with using CPAP mask versus stacked breathing on chest expansion and pulmonary function in patients with pneumonia .

Research hypothesis:- the investigators hypothesized that stacked breathing exercise is more effective on chest expansion and pulmonary function and more tolerant to patients with pneumonia than NIV with using CPAP mask.

Patients and methods Research design:- Quasi experimental research design will be utilized to fulfill the aim of this study.

Study variables:-

* The independent variables are NIV with using CPAP mask and stacked breathing exercise . -The dependent variables are the patients ' outcomes which include:-

  1. Chest expansion.
  2. Pulmonary functions.
  3. Duration of ICU stay.
  4. Complications as respiratory complications and general complications.
  5. Mortality rate.

     Research settings:

     The study will be conducted in 4 settings include:- Chest intensive care unit at Assiut university hospital. General intensive care unit at Assiut university hospital. Obstetric intensive care at women health hospital. Trauma intensive care unit at Assiut university hospital.

     Sample:- A convenience sample of 60 male and female adult patients will be taken, the patients will be classified into two equal groups , 30 patients for each group. CPAP mask group will receive NIV with using CPAP mask and stacked breathing group who will receive stacked breathing exercise.

     Tools of the study:- The following tools will be used to collect data for study:- Tool [1]:- patient assessment sheet which will be developed by the researcher and uses to monitor hemodynamic parameters, assessment of respiratory system, assessment of laboratory findings , fluid balance in addition to socio-demographic and medical data . It includes 5 parts:- Part (1): Socio-demographic and medical data as patient code , age , sex , past history

     , present illness, cause of admission , date of admission, date of discharge and length of ICU stay. This part also includes assessments of hemodynamic parameters system include (Mean arterial pressure (MAP), heart rate (HR), temperature and CVP readings) and laboratory findings every day.

     Part (3): Assessment of respiratory system which includes :-
* Chest condition as respiratory rate ,cough (dry or productive, strong or weak ), sputum characteristics: (amount , viscosity and color), dyspnea , orthopnea , pain with breathing and also assessment of sputum and blood culture.
* Auscultation of the chest for breathing sounds and determine if there are abnormal breathing e.g [wheezing, bronchospasm, crepitation .....] every shift.
* chest x-ray and ventilator profile.
* Assessment of chest expansion.
* Assessment of pulmonary functions Part (4): Fluid balance chart which include fluid intake and output. Part (5):Medication chart. Tool [2]: pneumonia treatment sheet which will be developed by researcher and uses to assess procedures done to the patient and includes 5 parts:- Part (1) : NIV with using CPAP mask. Part (2) : Stacked breathing exercise Tool [3]: Outcome evaluation sheet which will be developed by the researcher and uses to assess the effect of NIV with using CPAP mask and Stacked breathing on :-

  * Chest expansion .
  * Pulmonary functions.
  * Days of staying in ICU.
  * Complications such as pulmonary complications as pulmonary edema, bronchitis , pulmonary embolism , respiratory failure ...others and general complications as acute renal failure , liver failure , multiple organ failure or …..others.
  * Mortality rate.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 - 60 years.
* patients of both genders.
* patients diagnosed with pneumonia.

Exclusion Criteria:

* Orthopedic conditions.
* Malignant conditions.
* Cognitive impairments.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-08-30 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
change chest expansion to the normal range | for 7 days
  change chest expansion as chest expansion measures will be in the normal range and it is measured by measuring tape in CM before and after the procedure
change pulmonary functions to the normal values | for 7 days
  pulmonary functions will be assessed by bed side pulmonary function test as Schneider's match blowing test .

CONTACTS AND LOCATIONS:
Overall Officials: Amal A Mohamed, MD, Principal Investigator — Assiut University
Locations (1):
- Assiut University Hospitals, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD